CLINICAL TRIAL: NCT04840628
Title: The Relationship Between the Nreural Drive and Intrinsic Positive End-expiratory Pressure of the Chronic Obstructive Pulmonary Disease Patients With Respiratory Failure
Brief Title: The Relationship Between the Neural Drive and Intrinsic Positive End-expiratory Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhang Jianheng, Clinical Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: YLS2020(142)
Record Dates: First submitted 2020-11-27; First posted 2021-04-12 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: neural respiratory drive; Intrinsic Positive End-expiratory Pressure; Chronic Obstructive Pulmonary Disease Patients
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: the chronic obstructive pulmonary disease patients with respiratory failure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neural respiratory drive (Experimental): neural respiratory drive assessed by EMGdi recorded from a multipair esophageal electrode
  Interventions: Other: Resistance of the respiratory system

INTERVENTIONS:
Other: Resistance of the respiratory system — increase the resistance of the respiratory system of the chronic obstructive pulmonary disease patients

SUMMARY:
To investigate the relation the nreural drive and intrinsic positive end-expiratory pressure(PEEPi) of the chronic obstructive pulmonary disease(COPD) patients with respiratory failure.In present study the PEEPi of COPD patients was increased by increasing the resistance of the respiratory system, the change of the neural drive was recorded.

DETAILED DESCRIPTION:
To investigate the relation the nreural drive and intrinsic positive end-expiratory pressure(PEEPi) of the chronic obstructive pulmonary disease(COPD) patients with respiratory failure.The diaphragm electromyogram (EMGdi) represents the neural drive to the diaphragm.A multi-pair esophageal electrode catheter was used to record the EMGdi.The PEEPi was assessed by the by the balloon-catheter in the multi-pair esophageal electrode catheter. In present study the PEEPi of COPD patients was increased by increasing the resistance of the respiratory system, the change of the neural drive( EMGdi) was obtained from the a multi-pair esophageal electrode catheter All the signal recorded in the computer. The relation the nreural drive assessed by EMGdi and intrinsic positive end-expiratory pressure(PEEPi) would be analysed.

ELIGIBILITY:
Inclusion Criteria:

chronic obstructive pulmonary disease patients with respiratory failure

Exclusion Criteria:

1. Heart failure
2. cardiac dysrhythmia
3. Loss of consciousness

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-07-03 (Actual)

PRIMARY OUTCOMES:
neural respiratory drive assessed by the root mean square of diaphragm electromyogram (EMGdi) of the chronic obstructive pulmonary disease patients with respiratory failure | 1 hour
  neural respiratory drive assessed by the root mean square of diaphragm electromyogram (EMGdi) obtained from the a multi-pair esophageal electrode catheter

CONTACTS AND LOCATIONS:
Locations (1):
- 1State Key Laboratory of Respiratory Disease, National clinical research center for respiratory disease, Guangzhou Institute of respiratory health. 2The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
we will share our data by publishing the paper